CLINICAL TRIAL: NCT05856474
Title: Surgical Management of Traumatic Pancreas Transection
Brief Title: Management of Traumatic Pancreas Transection
Status: Recruiting | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: pancreas transection; A-ER-110-209 (Other: National Cheng Kung University Hospital)
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Pancreatectomy
MeSH Terms: interventions — Pancreatectomy; Pancreaticojejunostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pancreatectomy — pancreaserving surgery, using end to side or end to end, pancreaticojejunostomy
  Other Names: pancreaticojejunostomy

SUMMARY:
The goal of this observational study is to learn about the type of surgical effect on pancreas transection.

The main questions aims to answer are:

* 1. does pancreas preserving able to decrease incidence of postoperative diabeters
* 2. what is cause of major cause of postoperative morbidity and mortality in pancreas transection

DETAILED DESCRIPTION:
The study design was a retrospective chart review and analysis of Traumatic Pancreas Transection(TPT) patients treated at National Cheng Kung University Hospital. The clinical records, including demographic data, computed tomographic location of pancreas transection with intraoperative confirmation of the pancreatic injury, associated intra-abdominal injuries, interval time between injury and operation, surgical procedure, presence of complication (pancreas and non pancreas related), timing of drain removal, duration of hospital stay and mortality recorded. The secondary end point of morbidity was assessed using the Clavien-Dindo classification.

Initial resuscitation was implemented using ATLS guide-lines. Damage-control laparotomy was applied in critically hemodynamic unstable patients.

In a relatively stable patient, damage control procedure using TAE to control solid organ ongoing hemorrhage and blood transfusion prior to pancreas and associated gastrointestinal surgery. Depending the surgeon preference, TPT patient underwent open or laparoscopic surgery, either using distal pancreatectomy, with or without splenectomy or pancreas preserving pancreatojejunostomy.

Early pancreas surgery is defined as undergoing pancreas reconstructive surgery within 48 hrs. while delayed is considered when beyond 48 hrs. Operative intervention in 42 each patient was individualized based on the surgeon's. Negative suction drain, using Jackson Pratt drain is placed just near proximal pancreas stump.

Drain was removed when the amount was less than 50 cc/day with or without drain amylase/lipase level is less than 3 times of normal serum level.

Morbidity was documented as systemic, intra-abdominal, or specific complications related directly to the pancreatic injury.

Mortality was defined as any cause of death during hospital days. All available postoperative data including blood glucose, Hb1AC, serum and drain amylase lipase level, timing of drain removal, morbidity, hospital stays and mortality was collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed to have pancreas injury confirmed to pancreas injury by laparotomy.

Exclusion Criteria:

* negative pancreas injury by laparotomy

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospital admission and underwent surgerical laparotomy in a single institution
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
post opereative diabetes | 6 month
  occurence of diabetes following pancreas resection and pancreas preserving surgery

SECONDARY OUTCOMES:
post removal drain outcome | 2 week to 4 weeks
  pseudocyst and abscess complication following drain removal

CONTACTS AND LOCATIONS:
Overall Officials: Yen- Shen Shan, Study Chair — National Cheng Kung University, College of Medicine
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
share data result finding in short term of incidence of post operative diabetes following distal pancreatectomy

REFERENCES:
- [Result] Saisho Y, Butler AE, Meier JJ, Monchamp T, Allen-Auerbach M, Rizza RA, Butler PC. Pancreas volumes in humans from birth to age one hundred taking into account sex, obesity, and presence of type-2 diabetes. Clin Anat. 2007 Nov;20(8):933-42. doi: 10.1002/ca.20543. PMID 17879305
- [Result] Krige JE, Jonas E, Thomson SR, Kotze UK, Setshedi M, Navsaria PH, Nicol AJ. Resection of complex pancreatic injuries: Benchmarking postoperative complications using the Accordion classification. World J Gastrointest Surg. 2017 Mar 27;9(3):82-91. doi: 10.4240/wjgs.v9.i3.82. PMID 28396721
- [Result] Bozdag Z, Kapan M, Ulger BV, Turkoglu A, Uslukaya O, Oguz A, Aldemir M. Factors affecting morbidity and mortality in pancreatic injuries. Eur J Trauma Emerg Surg. 2016 Apr;42(2):231-5. doi: 10.1007/s00068-015-0526-8. Epub 2015 Apr 8. PMID 26038044